CLINICAL TRIAL: NCT02966340
Title: Repurposing alpha1 Noradrenergic Antagonists for Alcoholism Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: 2014-0966; F31AA022845-01 (NIH); Kaye2 (Other: Study Team)
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Alcoholism
Keywords: Alcoholism; Prazosin; Startle Potentiation; Norepinephrine; Anxiety; Fear; Stress
MeSH Terms: conditions — Alcoholism; Anxiety Disorders | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prazosin 1st visit, Placebo 2nd visit (Experimental): All participants receive 2mg prazosin and placebo in a cross-over design (e.g., one pill per visit). The order of prazosin vs placebo is counterbalanced between subjects (e.g., half participants receive prazosin at study visit 1 and half participants receive placebo at study visit 1).
  Interventions: Drug: Prazosin; Drug: Placebo
- Placebo 1st visit, Prazosin 2nd visit (Experimental): All participants receive 2mg prazosin and placebo in a cross-over design (e.g., one pill per visit). The order of prazosin vs placebo is counterbalanced between subjects (e.g., half participants receive prazosin at study visit 1 and half participants receive placebo at study visit 1).
  Interventions: Drug: Prazosin; Drug: Placebo

INTERVENTIONS:
Drug: Prazosin — 2mg Prazosin
Drug: Placebo — Placebo

SUMMARY:
Double-blind, placebo-controlled, cross-over design study examining the effects of a norepinephrine alpha1 receptor antagonist (prazosin) on stress reactivity in a laboratory stressor task.

DETAILED DESCRIPTION:
OBJECTIVES

The first objective of the current study is to examine norepinephrine alpha1 (NE-alpha1) receptor involvement in reactivity to unpredictable stressors in humans, by using the NPU stress task in conjunction with an alpha1-blocker, prazosin. The second objective of the study is to provide preliminary evidence that prazosin is effective at reducing stress-reactivity in alcoholics in early abstinence.

PARTICIPANTS

Sixty-four healthy adult participants and sixty-four participants with an Alcohol Use Disorder in early abstinence.

STUDY OVERVIEW

Sixty-four healthy adult participants (32 males & 32 females) will be recruited to participate in a double-blind, placebo-controlled, cross-over design study examining the effects of a NE-alpha1 antagonist (prazosin) on the defensive (physiological and self-report affect) response to stressors using a well-validated animal-human translational stressor task. Participants will complete two overnight study visits where 2 mg prazosin and placebo are administered on separate visits separated by approximately 7 days. Drug order is randomly assigned and counterbalanced across participants (double-blind; study visits 1-2). On each of these two study visits, participants will complete the No Shock, Predictable Shock, Unpredictable Shock (NPU) task 90 minutes after drug administration. The NPU task is designed to examine stress reactivity to predictable and unpredictable stressors (i.e., electric shock). These two visits provide for a within-subject evaluation of the effect of acute antagonism of alpha1-NE receptors (via prazosin) to investigate the role of this NE mechanism in unpredictable (vs. predictable) stressor response.

After the full healthy adult/control sample has completed the study, the investigators will conduct preliminary data analysis to evaluate the first study hypothesis. These analyses are used to evaluate the sensitivity of the NPU task to NE-alpha1 mechanisms and its potential utility as an early surrogate endpoint for stress-related relapse mechanisms in alcoholism. The investigators will only recruit the sample of sixty-four alcoholic participants to complete the study if the first hypothesis is initially supported with healthy controls. These participants will meet Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) criteria for Alcohol Use Disorder (at least moderate severity) and be in early abstinence (1-8 weeks). All other study procedures will be identical for this sample.

OUTCOME MEASURES

The primary outcome is startle potentiation during the NPU task and the secondary outcome is self-reported retrospective fear/anxiety during the NPU task.

HYPOTHESES

1. Prazosin (2mg vs. placebo) will reduce stress reactivity to unpredictable (vs. predictable) stressors measured via startle potentiation and self-report.
2. Abstinent alcoholics (vs. controls) will display elevated stress reactivity to unpredictable (vs. predictable) stressors measured via startle potentiation and self-report.
3. The predicted effects of prazosin on reducing stress reactivity to unpredictable (vs. predictable) stressors (Hypothesis 1) measured via startle potentiation and self-report will be moderated by alcoholism, such that the effects of prazosin will be larger in abstinent alcoholics than control participants.

ELIGIBILITY:
INCLUSION CRITERIA: All Participants

* Can read and write in English.
* Ages of 18-50 years.

INCLUSION CRITERIA: Control Participants

* No current or lifetime history of Substance Use Disorder (except tobacco).

INCLUSION CRITERIA: Alcoholic Participants

* Current Alcohol Use Disorder with 1-8 weeks completely free from alcohol consumption.

Exclusion criteria are divided into three broad categories of Medical, Psychiatric/Behavioral, and Medications/Therapies.

EXCLUSION CRITERIA: Medical

* Colorblind
* Blood alcohol concentration (BAC) > 0.00
* Systolic BP <100 after five minutes seated.
* Systolic BP drop >20 mmHg after two minutes standing.
* Systolic BP drop >10 mgHg AND report dizziness, lightheadedness, unsteadiness or other problems (e.g, nausea, blurry vision) after two minutes standing.
* Heart rate >100 beats/ minute after two minutes seated.
* Heart rate <60 beats/ minute after two minutes seated.
* Scheduled for cataract surgery prior to study completion.
* Past or current coronary artery disease, cerebrovascular accident, congestive heart failure.
* Current renal insufficiency, liver insufficiency, pancreatitis, immunosuppressive therapy, or cancer with systemic effects or therapy.
* Benign positional vertigo, Meniere's disease or narcolepsy
* Current diabetes or polyneuropathy
* Previous allergic or adverse reaction to prazosin or other alpha1 norepinephrine antagonist.
* Other self-reported acute or unstable illness that, in the opinion of the study team, would preclude a safe and reliable study participation.

EXCLUSION CRITERIA: Female Participants Only

* Non-negative urine pregnancy test.
* Women of childbearing potential (see definition below) must agree to use one of the following forms of birth control until after study completion. Acceptable birth control is defined as the following methods of contraception: abstinence; hormonal contraceptives (e.g. combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device (IUD) or intrauterine system (IUS); vasectomy of partner and tubal ligation; "single" barrier methods of contraception (e.g. male condom, female condom, cervical cap, diaphragm, contraceptive sponge) with use of spermicide; or "double barrier" method of contraception (e.g. male condom with diaphragm, male condom with cervical cap).
* Breastfeeding

NOTE: Women of childbearing potential are females who have experienced menarche and do not meet the criteria for women not of childbearing potential. Women not of childbearing potential are females who are permanently sterile (e.g., hysterectomy, bilateral oophorectomy) or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause.

EXCLUSION CRITERIA: Psychological/Behavioral Exclusion

* Self-reported lifetime diagnosis of schizophrenia, schizoaffective disorder, psychotic disorder not otherwise specified (NOS), bipolar disorder, borderline personality disorder, or any neurocognitive disorder.

EXCLUSION CRITERIA: Medications/Therapies

* Currently prescribed or used within 72 hours: prazosin or other alpha1-NE antagonist (e.g., doxazosin, terazosin).
* Previous adequate trial of prazosin for alcohol use disorder or PTSD.
* Currently prescribed or used within 72 hours: Stimulants (e.g., d-amphetamine, methylphenidate) or alternative medications with stimulant properties (e.g., ephedra, pseudoephedrine).
* Currently prescribed or used within 72 hours: Sildenafil (Viagra), tadalafil (Cialis), or vardenafil (Levitra).
* Currently prescribed or used within 72 hours: beta-blockers (e.g., propranolol), alpha2 agonists (e.g., clonidine, guanfacine), or Serotonin-norepinephrine reuptake inhibitor (SNRI) anti-depressants (e.g., venlafaxine, duloxetine).
* Currently used daily or used within 72 hours: alpha1 agonists (e.g., midodrine, metaraminol, oxymetazoline, phenylephrine).
* Currently used daily or used within 72 hours: Benzodiazepines (e.g., diazepam, chlordiazepoxide, lorazepam, clonazepam, alprazolam), zolpidem (Ambien), zaleplon (Sonata), zopiclone (Imovane), eszopiclone (Lunesta), doxepin (Silenor).
* Currently prescribed and used daily or used within 72 hours: Trazodone (males only)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Curtin, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share on Open Science Framework de-identified and anonymous physiology (e.g., Electromyography (EMG) startle response) and self-report survey/questionnaire data collected from participants during the study.

REFERENCES:
- See also: Dr. John Curtin's Addiction Research Center — http://dionysus.psych.wisc.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In order to enroll 64 participants with valid data, 70 participants were randomized to account for 4 lost early in study flow (one data collection error, two startle non-responders, and one withdrawn after visit 1).
Period: Overall Study
Arm/Group | Prazosin 1st Visit, Placebo 2nd Visit | Placebo 1st Visit, Prazosin 2nd Visit
Started | 37 | 33
Completed | 34 | 30
Not Completed | 3 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — data acquisition error | 1 | 0
Not completed — startle non-responder | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants Who Completed the Study: All participants receive 2mg prazosin and placebo in a cross-over design (e.g., one pill per visit). The order of prazosin vs placebo is counterbalanced between subjects (e.g., half participants receive prazosin at study visit 1 and half participants receive placebo at study visit 1).
  Results are to be reported by treatment (placebo vs prazosin) each of which include results for all participants. Therefore we report baseline characteristics for the entire group.
Arm/Group | All Participants Who Completed the Study
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 64
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 59
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 41
  More than one race | 6
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: Startle Potentiation During Stress Reactivity Task.
Description: The unpredictable shock and predictable shock startle response potentiation (vs. no shock) during the administration of the NPU stressor task. Values represent point estimate of effect from unadjusted general linear model analyses with 95% confidence intervals
Time Frame: 7 days
Measure: Mean (95% Confidence Interval); unit: startle potentiation (μV)
Groups:
- Prazosin 2mg Trials; Placebo Trials: All participants receive 2mg prazosin and placebo in a cross-over design (e.g., one pill per visit). The order of prazosin vs placebo is counterbalanced between subjects (e.g., half participants receive prazosin at study visit 1 and half participants receive placebo at study visit 1).
  Prazosin: 2mg Prazosin
  Placebo: Placebo
Arm/Group | Prazosin 2mg Trials | Placebo Trials
Number analyzed (Participants) | 64 | 64
startle potentiation (μV)
  Predictable Shock | 45.7 [33.5 to 57.8] | 40.1 [29.7 to 50.4]
  Unpredictable Shock | 33.2 [24.3 to 42.1] | 25.2 [16.6 to 33.8]

2. Secondary Outcome: Self-reported Anxiety Potentiation During Stress Reactivity Task.
Description: After the No-shock, Predictable-shock, Unpredictable-shock (NPU) task participants retrospectively reported their anxiety/fear during each condition on a 5-point likert scale (1 = 'Not at all anxious/ fearful', 5 = 'Very anxious/fearful'). The startle response is a defensive reflex that is elicited by an auditory stimuli (e.g., 50ms white noise) and measured via eyeblink electromyogram (EMG) activity over the obicularis oculi muscle. Startle potentiation is calculated as the increase in startle during unpredictable and predictable stressors relative to a no-stressor condition in the NPU task. Outcome is anxiety potentiation during unpredictable shock and predictable shock (vs. no-shock) conditions. This was assessed with a single question, total possible range was 1-5.
Time Frame: 7 days
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Prazosin 2mg Trials | Placebo Trials
Number analyzed (Participants) | 64 | 64
units on a scale
  Predictable Shock | 2.0 [1.7 to 2.3] | 2.1 [1.8 to 2.4]
  Unpredictable Shock | 2.3 [2.0 to 2.6] | 2.4 [2.1 to 2.7]

ADVERSE EVENTS:
Time Frame: Up to 24 hours
Description: Nurses completed Adverse Events (AE) evaluations at 1, 3, 4, 5, and 6 hours post-dose at each study visit.
Arm/Group | Prazosin 2mg Trials | Placebo Trials
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/64
Other Adverse Events (participants affected / at risk) | 30/64 | 3/64
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prazosin 2mg Trials (N=64) | Placebo Trials (N=64)
Dizzyness (Vascular disorders) | 16 (16) | 0 (0)
Lightheadedness (Vascular disorders) | 12 (12) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 0 (0)
Headache (Vascular disorders) | 3 (3) | 1 (1)
Drowsiness (Vascular disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT02966340/Prot_SAP_000.pdf